CLINICAL TRIAL: NCT04323761
Title: Expanded Access Treatment Protocol: Remdesivir (RDV; GS-5734) for the Treatment of SARS-CoV2 (CoV) Infection
Brief Title: Expanded Access Treatment Protocol: Remdesivir (RDV; GS-5734) for the Treatment of SARS-CoV2 (CoV) Infection (COVID-19)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-540-5821; 2020-001453-49 (EudraCT Number)
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Remdesivir — Intravenous infusion administered over a 30 to 120 minute period
  Other Names: GS-5734™; Veklury®

SUMMARY:
The primary objective of this study is to provide expanded access of remdesivir (RDV) for the treatment of severe acute respiratory syndrome coronavirus (SARS-CoV2) infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants ≥ 18 years of age), or willing and able to provide assent (participants ≥ 12 and < 18 years of age, where locally and nationally approved) prior to performing study procedures. For participants ≥ 12 and < 18 years of age, a parent or legal guardian willing and able to provide written informed consent prior to performing study procedures.
* Age ≥ 18 years or aged ≥ 12 and < 18 years of age weighing ≥ 40 kg (where permitted according to local law and approved nationally and by the relevant institutional review board (IRB) or independent ethics committee (IEC))
* Hospitalized with confirmed SARS-CoV2 by polymerase chain reaction (PCR) or known contact of confirmed case with syndrome consistent with coronavirus disease (COVID-19) with PCR pending
* Oxygen saturation (SpO2) ≤ 94% on room air or requiring supplemental oxygen at baseline
* Alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN) by local laboratory measure and/or ALT < 3 x ULN and bilirubin < 2 x ULN
* Females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Lactating females must agree to discontinue nursing before the study drug is administered and while they are participating in the study

Exclusion Criteria:

* Evidence of multiorgan failure including but not limited to coagulopathy (significant thrombocytopenia), hepatic failure (elevated bilirubin) or renal failure (low urine output or estimated glomerular filtration rate (eGFR) < 30 mL/min), or significant cardiomyopathy (low cardiac output)
* Use of more than 1 pressor for septic shock (note that use of 1 pressor at low/medium doses for inotropic support due to the use of sedation and paralytics while on the ventilator is allowed)
* Renal failure (eGRF < 30 mL/min using the Cockcroft-Gault formula for participants ≥ 18 years of age and Schwartz Formula for participants < 18 years of age) or dialysis or continuous Veno-Venous Hemofiltration)
* Eligible for enrollment in a randomized clinical trial studying remdesivir for treatment of SARS-CoV2 at the medical facility where the participant is admitted
* Known hypersensitivity to the study drug, the metabolites, or formulation excipient
* Requiring venous arterial (V-A) extracorporeal membrane oxygen (ECMO) (venous venous (V-V) ECMO is not an exclusion criteria)

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (272):
- United States (165):
  - University of Alabama- Birmingham, Birmingham, Alabama
  - Banner- University Medical Center Phoenix, Phoenix, Arizona
  - Community Regional Medical Centers (CRMC), Fresno, California
  - St. Jude Medical Center, Fullerton, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Huntington Hospital, Pasadena, California
  - Scripps Mercy Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, Medical Center (Parnassus Campus), San Francisco, California
  - Regional Medical Center, San Jose, California
  - San Mateo Medical Center, San Mateo, California
  - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - PIH Health Whittier Hospital, Whittier, California
  - The Medical Center Of Aurora, Aurora, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Middlesex Health, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - The Stamford Health Medical Group- Pulmonary Associates, Stamford, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Aventura Hospital and Medical Center, Aventura, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Investigational Drug Services, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Wellstar Atlanta Medical Center, Atlanta, Georgia
  - Piedmont Columbus Regional-Midtown Hospital, Columbus, Georgia
  - Grady Health System- Grady Memorial Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Swedish Hospital, Chicago, Illinois
  - Mercy Hospital & Medical Center, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - St. Vincent Hospital and Health Care Center, Inc., Carmel, Indiana
  - Richard L Roudebush Indianapolis VA, Indianapolis, Indiana
  - Riverview Health, Noblesville, Indiana
  - Our Lady of the Lakes Regional Medical Center, Baton Rouge, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Slidell Memorial Hospital, Slidell, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - CalvertHealth Medical Center, Prince Frederick, Maryland
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Steward St. Elizabeth's Medical Center of Boston, Inc., Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Lawrence General Hospital, Lawrence, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Wayne Statue University/ Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Health Care Corporation, Flint, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - CarePoint Health Bayonne Medical Center, Bayonne, New Jersey
  - Clara Maass Medical Center, Belleville, New Jersey
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack Meridian Health - JFK Medical Center, Edison, New Jersey
  - Trinitas Regional Medical Center, Elizabeth, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Robert Wood Johnson University Hospital Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Christ Hospital- Carepoint Health, Jersey City, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Atlantic Health System/ Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - Ocean Medical Center, Oakhurst, New Jersey
  - Bayshore Medical Center, Red Bank, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Atlantic Health System/Overlook Medical Center, Summit, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Capital Health, Trenton, New Jersey
  - Virtua Health Voorhees Campus, Voorhees Township, New Jersey
  - St. Peter's Hospital, Albany, New York
  - Mount Sinai Queens, Astoria, New York
  - Good Samaritan Hospital Medical Center, Bay Shore, New York
  - Southside Hospital, Bay Shore, New York
  - The Brooklyn Hospital Center, Brooklyn, New York
  - Kingsbrook Jewish Medical Center, Brooklyn, New York
  - University Hospital Brooklyn (SUNY Downstate), Brooklyn, New York
  - Woodhull Medical Center, Brooklyn, New York
  - Kings County Hospital Center, Brooklyn, New York
  - New York Harbor VA Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Interfaith Medical Center, Brooklyn, New York
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Mount Sinai Brooklyn, Brooklyn, New York
  - New York City Health and Hospitals - Coney Island, Brooklyn, New York
  - Kaleida Health System, Buffalo, New York
  - Nassau University Medical Center, East Meadow, New York
  - New York Presbyterian- Queens, Flushing, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - New York City Health and New York City Health and Hospitals - Metropolitan- Metropolitan, New York, New York
  - NewYork-Presyterian/Columbia University Irving Medical Center- Milstein Hospital, New York, New York
  - New York City Health + Hospitals / Harlem, New York, New York
  - New York Presbyterian Lower Manhattan Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai South Nassau, Oceanside, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Ellis Hospital, Schenectady, New York
  - Staten Island University Hospital- Northwell Health (North Campus), Staten Island, New York
  - Stony Brook University Hospital/ Stony Brook Children's, Stony Brook, New York
  - Lincoln Medical Center, The Bronx, New York
  - St Barnabus Hospital, The Bronx, New York
  - Montefiore Medical Center, Weiler Campus, The Bronx, New York
  - Montefiore Health System Moses Medical Center, The Bronx, New York
  - Samaritan Hospital, Troy, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Atrium Health- Carolinas Medical Center, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Francis Hospital, Tulsa, Oklahoma
  - St. Luke's Hospital - Bethlehem Campus, Bethlehem, Pennsylvania
  - Mercy Catholic Medical Center - Fitzgerald Campus, Darby, Pennsylvania
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - St. Francis Hospital, Greenville, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Texas Department of Criminal Justice Hospital (Hospital Galveston)/University of Texas Medical Branch, Galveston, Texas
  - HCA Houston Healthcare West, Houston, Texas
  - Covenant Medical Center, Lubbock, Texas
  - Methodist Mansfield Medical Center, Mansfield, Texas
  - Methodist Healthcare System of San Antonio, Ltd. LLP, dha, Methodist Hospital, San Antonio, Texas
  - Saint Mark's Hospital, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Henrico Doctors Hospital, Richmond, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - University of Washington Medical Center- Montlake Campus, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Gold Coast Hospital, Southport
- Austria (5):
  - Landeskrankenhaus Graz West, Graz
  - Universitätsklinik für Innere Medizin II, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - Sozialmedizinisches Zentrum Süd - Kaiser-Franz-Josef-Spital, Vienna
  - Medical University and General Hospital Vienna, Vienna
- Belgium (7):
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Hôpital Civil Marie Curie, Lodelinsart
- Canada (2):
  - William Osler Health System, Brampton, Ontario
  - The Ottowa Hospital, Ottawa, Ontario
- Nicosia General Hospital, Nicosia, Cyprus
- Czechia (3):
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Eticka komise pro multicentircke klinicke hodnoceni Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce, Praha 8 - Liben
- Rigshospitalet, Copenhagen, Denmark
- Estonia (2):
  - Põhja-Eesti Regionaalhaigla, Tallinn
  - Vilnius University, Tartu
- France (10):
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Regional Universitaire Brest Hôpital de la Cavale Blanche à Brest, Brest
  - Centre Hospitalier Universitaire Gabriel-Montpied, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôpital Raymond Poincaré, Garches
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Charles-Nicolle, Rouen
  - Hôpital Purpan, Toulouse
- Germany (10):
  - Saint Josef Hospital Ruhr Universitaet Bochum, Bochum
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitatsklinikum, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Caritas-Krankenhaus St. Josef, Regensburg
  - Klinikum Würzburg Mitte, Würzburg
- Greece (2):
  - University General Hospital of Patras Panagia I Voithia, Pátrai
  - General Hospital of Thessaloniki George Papanikolaou, Thessaloniki
- Kenézy Gyula Kórház És Rendelőintézet, Debrecen, Hungary
- Landspítali, Reykjavik, Iceland
- Kerry University Hospital, Tralee, Ireland
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Hasharon Hospital, Petah Tikva
  - Sheba Medical Center at Tel Hashomer, Ramat Gan
- Italy (13):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico di Bari, Bari
  - Azienda Ospedaliero Universitaria, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Presidio Ospedaliero Garibaldi-Nesima, Catania
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale San Gerardo di Monza, Monza
  - Azienda Ospedaliera dei Colli, Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS Istituto Nazionale per le Malattie Infettive Lazzaro Spallanzani, Roma
  - Azienda Ospedaliero Universitaria, Turin
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Vilnius University, Vilnius
- Netherlands (2):
  - Radboud Universitair Medisch Centrum, Nijmegen
  - HagaZiekenhuis, The Hague
- Poland (4):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewódzki Specjalistyczny Szpital im. dr. Wł. Biegańskiego, Lodz
  - Wielospecjalistyczny Szpital Miejski Im Józefa Strusia Zakład Opiekuńczo Leczniczy, Poznan
  - Wojewódzki Szpital Specjalistyczny Megrez Sp. z o.o., Tychy
- Portugal (4):
  - Centro Hospitalar Universitário de Lisboa Central - Hospital Curry Cabral, Lisbon
  - Centro Hospitalar Universitário do Porto E.P.E., Porto
  - Centro Hospitalar Universitário De São João, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia
- Romania (3):
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals, Bucharest
  - Spitalul Clinic de Boli Infecţioase Sfânta Parascheva Iaşi, Iași
  - Clinical hospital for infectious disease, Timișoara
- Univerzitná Nemocnica L. Pasteura Košice - Pracovisko Rastislavova 43, Košice, Slovakia
- Slovenia (2):
  - Univerzitetni Klinicni Center Ljubljana, Ljubljana
  - Univerzitetni Klinicni Center Maribor, Maribor
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Virgen De La Salud, Santa Cruz de Tenerife
  - Hospital Virgen De La Salud, Toledo
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (7):
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubünden, Chur
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Hôpital du Valais -Hôpital de Sion, Sion
- United Kingdom (5):
  - University Hospital of Wales, Cardiff and Vale NHS Trust, Cardiff
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - St. George's Hospital, London
  - Southampton University Hospital, Southampton